CLINICAL TRIAL: NCT00147654
Title: A Randomized, Double Blind, Placebo Controlled, Four Arm (Placebo, Tolterodine ER, Tamsulosin, and Tolterodine ER Plus Tamsulosin) Study To Evaluate The Clinical Efficacy And Safety Of Tolterodine ER 4 mg In Men Who Have Frequency and Urgency, With Or Without Urinary Urge Incontinence, With Or Without Bladder Outlet Obstruction
Brief Title: Effect and Safety Of Detrol LA In Men With Overactive Bladder Symptoms With Or Without Bladder Outlet Obstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6121120
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Tolterodine Tartrate; Tamsulosin

INTERVENTIONS:
Drug: Tolterodine ER 4 mg QD
Drug: Tamsulosin 0.4 mg QD

SUMMARY:
The primary objective of the trial is to evaluate the effect of tolterodine ER plus tamsulosin versus placebo on patient perception of overall treatment benefit in men who have frequency and urgency, with or without urinary urge incontinence (UUI), with or without bladder outlet obstruction (BOO).

ELIGIBILITY:
Inclusion Criteria:

* Male 40 years of age
* Clinical signs and symptoms of frequency and urgency, with or without UUI, with or without BOO, for at least three months
* Mean urinary frequency of 8 micturitions/24h verified by the Screening micturition diary

Exclusion Criteria:

* Post-void residual urine volume (PVR) of > 200 ml as measured by an ultrasound
* Maximum urinary flow rate (Qmax) of < 5 ml/second as measured by a flowmeter; a voided volume of 75 ml is required in order to accurately record the Qmax
* Prescribed and administered an antimuscarinic or antispasmodic within 1 month
* Prescribed and administered an a-1-adrenergic antagonist within 2 weeks

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830
Dates: Start 2004-11; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Patient Perception of Treatment Benefit at Week 12:
Treatment benefit, treatment satisfaction, and willingness to continue treatment questions at week 12

SECONDARY OUTCOMES:
Micturition Diary- Change in number of urge incontinence episodes per 24 hours at week 1, week 6 and 12 relative to baseline.
Change in number of urge episodes per 24 hours at week 1, week 6 and 12 relative to baseline.
Change in number of micturitions per 24 hours at week 1, week 6 and 12 relative to baseline.
Change in number of daytime micturitions per 24 hours at week 1, week 6 and 12 relative to baseline
Change in number of nighttime micturitions per 24 hours at week 1, week 6 and 12 relative to baseline
Change in the average severity of the Urinary Sensation Scale at week 1, week 6, and week 12 relative to baseline
Change in number of OAB micturition episodes per 24 hours (OAB micturition is defined as micturition episodes associated with Urinary Sensation Scale score 3) at week 1, week 6 and week 12 relative to baseline
Change in number of daytime OAB micturition episodes per 24 hours (OAB micturition is defined as micturition episodes associated with Urinary Sensation Scale score 3) at week 1, week 6 and week 12 relative to baseline
Change in number of nighttime OAB micturition episodes per 24 hours. (severe OAB micturition is defined as micturition episodes associated with Urinary Sensation Scale score 4) at week 1, week 6 and week 12 relative to baseline
Change in number of severe OAB micturition episodes per 24 hours (severe OAB micturition is defined as micturition episodes associated with Urinary Sensation Scale score 4) at week 1, week 6 and week 12 relative to baseline
Change in number of daytime severe OAB micturition episodes per 24 hours (severe OAB micturition is defined as micturition episodes associated with Urinary Sensation Scale score 4) at week 1, week 6 and week 12 relative to baseline
Change in number of nighttime severe OAB micturition episodes per 24 hours (severe OAB micturition is defined as micturition episodes associated with Urinary Sensation Scale score 4) at week 1, week 6 and week 12 relative to baseline
International Prostate Symptom Score (I-PSS):
Change in I-PSS total score at weeks 1, 6 and 12 relative to baseline
Change in I-PSS individual item scores (Q1, Q2, Q3, Q4, Q5, Q6, and Q7) at weeks 1, 6 and 12 relative to baseline
Change in I-PSS irritative domain (Sum of Q2, Q4, and Q7) at weeks 1, 6 and 12 relative to baseline
Change in I-PSS obstructive domain (Sum of Q1, Q3, Q5, and Q6) at weeks 1, 6 and 12 relative to baseline
Change in I-PSS index score (Sum Q1 to Q7) at weeks 1, 6 and 12 relative to baseline
Change in I-PSS QoL score (Q8) at weeks 1, 6 and 12 relative to baseline
Patient perception of urgency:
Change in the Perception of Urgency Scale (3 point scale) at week 1, week 6 and week 12 relative to baseline
Change in Patient's Perception of Bladder Condition at week 1, week 6 and week 12 relative to baseline
Patient Perception of Treatment benefit at week 1 and week 6
Treatment benefit and treatment satisfaction questions will be completed at week 1 and week 6
Change in International Continence Society Male (ICSmaleLF) Questionnaire (long form modified) individual item scores at Week 1, Week 6 and Week 12 relative to baseline
Change in the total score of Overactive Bladder Questionnaire (OABq) and change in total scores for each domain of OABq at week 6 and week 12 relative to baseline
Change in the total score of International Index of Erectile Function (IIEF) and change in total scores for each domain of IIEF Questionnaire at week 6 and week 12 relative to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (95):
- United States (95):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Homewood, Alabama
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Culver City, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Murrieta, California
  - Pfizer Investigational Site, Poway, California
  - Pfizer Investigational Site, San Bernardino, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, New Britain, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, Wellington, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Columbus, Georgia
  - Pfizer Investigational Site, Roswell, Georgia
  - Pfizer Investigational Site, Melrose Park, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Brighton, Massachusetts
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, O'Fallon, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Missoula, Montana
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Cherry Hill, New Jersey
  - Pfizer Investigational Site, Edison, New Jersey
  - Pfizer Investigational Site, Hamilton, New Jersey
  - Pfizer Investigational Site, Lawrenceville, New Jersey
  - Pfizer Investigational Site, Marlton, New Jersey
  - Pfizer Investigational Site, Mount Laurel, New Jersey
  - Pfizer Investigational Site, Sewell, New Jersey
  - Pfizer Investigational Site, Voorhees Township, New Jersey
  - Pfizer Investigational Site, Westhampton, New Jersey
  - Pfizer Investigational Site, Woodbury, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Bay Shore, New York
  - Pfizer Investigational Site, Carmel, New York
  - Pfizer Investigational Site, Cortlandt Manor, New York
  - Pfizer Investigational Site, Garden City, New York
  - Pfizer Investigational Site, Manhasset, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Orchard Park, New York
  - Pfizer Investigational Site, Poughkeepsie, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Bala-Cynwyd, Pennsylvania
  - Pfizer Investigational Site, Bryn Mawr, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, State College, Pennsylvania
  - Pfizer Investigational Site, Wynnewood, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Greenwood, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Prosperity, South Carolina
  - Pfizer Investigational Site, Saluda, South Carolina
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Milan, Tennessee
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Provo, Utah
  - Pfizer Investigational Site, Alexandria, Virginia
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Fairfax, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Cheyenne, Wyoming

REFERENCES:
- [Derived] Kaplan SA, Roehrborn CG, Rovner ES, Carlsson M, Bavendam T, Guan Z. Tolterodine and tamsulosin for treatment of men with lower urinary tract symptoms and overactive bladder: a randomized controlled trial. JAMA. 2006 Nov 15;296(19):2319-28. doi: 10.1001/jama.296.19.2319. PMID 17105794
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6121120&StudyName=Effect+and+Safety+Of+Detrol+LA+In+Men+With+Overactive+Bladder+Symptoms+With+Or+Without+Bladder+Outlet+Obstruction